CLINICAL TRIAL: NCT00386581
Title: Phase III Multicenter, Randomized, Double-Blind Placebo-Controlled Outpatient Study of Efficacy, Tolerability, and Safety of Once-Daily Atomoxetine Hydrochloride Versus Placebo in Russian Children and Adolescents With Attention-Deficit/Hyperactivity Disorder
Brief Title: Efficacy, Tolerability, and Safety of Once-Daily Atomoxetine Hydrochloride Versus Placebo in Russian Children and Adolescents With Attention-Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9081; B4Z-MW-LYCZ
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: atomoxetine
Drug: placebo

SUMMARY:
The study is designed to investigate the acute treatment efficacy, safety, and tolerability of atomoxetine on a once-daily dosing strategy (in the morning). It incorporates a 6-week acute treatment period and a 2-week discontinuation phase. The assessments in this study include a standard assessment of ADHD symptomatology using a Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition™, investigator-administered rating scale.

ELIGIBILITY:
Inclusion Criteria

* Subjects must have ADHD that meets the DSM-IV criteria
* Aged 6 to 16 years.
* Subjects must not have taken any medication used to treat ADHD.
* Laboratory results must show no significant abnormalities
* Baseline ECG results must not show an abnormality
* Subjects must be able to swallow capsules.
* Subjects must be of normal intelligence.

Exclusion Criteria

* Weigh less than 20 kg or more than 60 kg at study entry.
* Subjects who, after an adequate trial with methylphenidate or amphetamine experience some benefit in ADHD signs and symptoms are excluded from participating.
* Have a history of Bipolar I or II disorder, psychosis, or PDD.
* Meet DSM-IV criteria for an anxiety disorder.
* Have a history of any seizure disorder.
* Patients at serious suicidal risk.
* Patients with narrow angle glaucoma
* Subjects who have a history of severe allergies .
* Have a history of alcohol or drug abuse within the past 3 months
* Screen positive for drugs of abuse not prescribed by a physician.
* Have cardiovascular disease and an increased heart rate and blood pressure.
* Have a medical condition that would increase sympathetic nervous system activity markedly or who are taking a medication on a daily basis.
* Have severe gastrointestinal narrowing
* Are during the study time likely to need psychotropic medications.
* Are likely to begin a structured psychotherapy aimed at ADHD symptoms.
* Have used a monoamine oxidase inhibitor (MAOI) during the 2 weeks
* Female subjects who are pregnant or who are breast-feeding.
* Are investigative site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study.
* Are, in the opinion of the investigator, unsuitable in any other way to participate in this study.
* Are employed by Lilly.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2004-07; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of atomoxetine administered as a single-daily dose with placebo in Russian children and adolescents with Attention-Deficit/Hyperactivity Disorder (ADHD).

SECONDARY OUTCOMES:
To compare improvement in symptoms associated with ADHD in children and adolescents achieved by once-daily dosing of atomoxetine or placebo, defined by a more than 25% reduction in the ADHDRS-IV-Parent:Inv total score and by mean reductions in Conners
To assess the safety and tolerability of once-daily dosing of atomoxetine in Russian children and adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow, Russia

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com